CLINICAL TRIAL: NCT01272245
Title: A Phase II Study of Omacetaxine (OM) and Low Dose Cytarabine (LDAC) in Older Patients With Acute Myelogenous Leukemia (AML) and High-Risk Myelodysplastic Syndrome (MDS)
Brief Title: Omacetaxine and Low Dose Cytarabine in Older Patients With Acute Myelogenous Leukemia (AML) and High-Risk Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0736; NCI-2013-02220 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Results first posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-04

CONDITIONS: Leukemia
Keywords: Acute Myelogenous Leukemia; AML; High-Risk Myelodysplastic Syndrome; MDS; Omacetaxine; Cytarabine; ARA-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Homoharringtonine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omacetaxine and Cytarabine (Experimental): Omacetaxine 1.25 mg/m2 SQ every 12 hours x 3 days + Cytarabine 20 mg SQ x 7 days of 4-7 week cycle.
  Interventions: Drug: Omacetaxine; Drug: Cytarabine

INTERVENTIONS:
Drug: Omacetaxine — 1.25 mg/m2 subcutaneously (SQ) every 12 hours (+/- 3 hours) for 3 days (Days 1-3). Each cycle will be 4-7 weeks.
Drug: Cytarabine — 20 mg subcutaneously every 12 hours (+/- 3 hours) for 7 days (Days 1-7). Each cycle will be 4-7 weeks.
  Other Names: ARA-C; Cytosar; Depo-Cyt; Cytosine Arabinosine Hydrochloride

SUMMARY:
The goal of this clinical research study is to learn if omacetaxine given with cytarabine can help to control the disease in patients with AML or high-risk MDS. The safety of the study drugs will also be studied.

DETAILED DESCRIPTION:
Study Drugs:

Omacetaxine is designed to block certain proteins, which may cause cancer cells to die.

Cytarabine is designed to insert itself into DNA (the genetic material of cells) of cancer cells and stop the DNA from repairing itself.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive omacetaxine and cytarabine as an injection under the skin. You will receive instructions on how to give these injections to yourself. You will be given a Research Medication Diary to record the drugs you take each day. You must bring the Research Medication Diary and any unused drugs with you to each study visit. You will also be told how to properly store the drugs.

On Days 1-3 of each cycle, you will give yourself an injection of omacetaxine every 12 hours (+/- 3 hours).

On Days 1-7 of each cycle, you will give yourself an injection of cytarabine every 12 hours (+/- 3 hours).

Each cycle will be 4-7 weeks, depending on how well the disease responds to the study drugs.

Depending on how the disease responds to the study drugs, the number of days you receive your injections may stay the same, increase, or decrease. Your doctor will discuss this with you.

Study Visits:

On Day 1 of each cycle, you will have a physical exam.

Women who are able to become pregnant must have a negative blood (about 1/2 teaspoon) or urine pregnancy test within 3 days before receiving the first dose of study drug.

Blood (about 1 tablespoon) will be drawn every week for routine tests. Once you have a response to treatment, blood will then be drawn every 2-4 weeks while you are receiving treatment. If your doctor thinks it is needed, you may have more blood samples drawn during Cycles 1 and 2.

On Day 21 of Cycle 1 (+/- 7 days), then every 4 weeks after that, you will have a bone marrow aspiration and/or biopsy to check the status of the disease. If the doctor thinks it is needed, these may be done more or less often, depending on your response to treatment.

Length of Study:

You may receive up to 24 cycles of treatment. You will be taken off study early if the disease gets worse or intolerable side effects occur.

Follow-up:

Once you stop taking the study drugs, you will have follow-up for 5 years.

Every 4-8 weeks, blood (about 1 tablespoon) will be drawn for routine tests. If you cannot return to the clinic, you may have blood drawn at a clinic close to your home.

Every 3-6 months, you will be contacted during a clinic visit and asked how you are doing. If you cannot make it to the clinic for this visit, you will be called. The phone call should last about 5 minutes.

This is an investigational study. Omacetaxine is FDA approved to treat patients with certain types of leukemia. Its use in this study is investigational. Cytarabine is FDA approved and commercially available for the treatment of AML. The use of these drugs in combination is investigational.

Up to 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Previously untreated AML (>/= 20% blasts). Patients with high-risk (intermediate-2 or high by International Prostate Symptom Score (IPSS) or ≥10% blasts) MDS will also be eligible. Prior therapy with hydroxyurea, biological or targeted therapy (e.g. flt3 inhibitors, other kinase inhibitors, azacitidine), or hematopoietic growth factors is allowed. A single or a two day dose of cytarabine (up to 3 g/m2) for emergency use is also allowed as prior therapy.
2. Age >/= 60 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status </= 2.
4. Adequate hepatic (serum total bilirubin </= 1.5 x ULN, serum glutamate pyruvate transaminase (SGPT) and/or serum glutamate oxaloacetate transaminase (SGOT) </= 2.5 x ULN) and renal function (creatinine </= 2.0 mg/dL).
5. Patients must be willing and able to review, understand, and provide written consent before starting therapy.

Exclusion Criteria:

1. New York Heart Association (NYHA) class III or IV heart disease, active ischemia or any other uncontrolled cardiac condition such as angina pectoris, clinically significant cardiac arrhythmia and requiring therapy, uncontrolled hypertension (blood pressure >/= 160 systolic and >/= 110 diastolic not responsive to antihypertensive medication), diabetes mellitus, or congestive heart failure.
2. Myocardial infarction in the previous 12 weeks (from the start of treatment).
3. Active and uncontrolled disease/infection as judged by the treating physician.
4. Pregnancy.
5. Acute promyelocytic leukemia (APL).
6. Women of childbearing potential and men who do not practice contraception. Non-childbearing is defined as >/= 1 year postmenopausal or surgically sterilized.
7. Women of childbearing potential and men must agree to use contraception prior to study entry and for the duration of study participation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Kantarjian, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 7/14/2011through 1/9/2015. All participants recruited at The University of Texas MD Anderson Cancer Center.
Groups:
- Omacetaxine and Cytarabine: Omacetaxine 1.25 mg/m2 subcutaneously (SQ) every 12 hours for 3 days + Cytarabine 20 mg SQ for 7 days of 4-7 week cycle.
Period: Overall Study
Arm/Group | Omacetaxine and Cytarabine
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Omacetaxine and Cytarabine
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 71 [60 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 19
Region of Enrollment [Number; unit: Count of Participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Remission (CR)
Description: Complete response (CR) defined as: Peripheral blood counts, no circulating blasts, neutrophil count ≥ 1.0 ×109/L, platelet count ≥ 100 ×109/L, bone marrow aspirate and biopsy, ≤5% blasts, no detectable auer rods, no extramedulary leukemia
Time Frame: Up to 4 months
Measure: Number; unit: percentage of participants
Arm/Group | Omacetaxine and Cytarabine
Number analyzed (Participants) | 36
percentage of participants | 44

2. Secondary Outcome: Evaluation of CR Duration
Description: The date of Complete Response to the date of loss of response or last follow-up.
Time Frame: Up to 5 years after completion of active treatment and while on study. Participants may receive up to 24 courses of study medication.
Measure: Median (Full Range); unit: Months
Arm/Group | Omacetaxine and Cytarabine
Number analyzed (Participants) | 16
Months | 10.6 [1.5 to 64.7]

3. Secondary Outcome: Disease-free Survival
Description: Time from date of treatment start until the date of first objective documentation of disease-relapse.
Time Frame: as for outcome 2
Measure: Median (Full Range); unit: Months
Arm/Group | Omacetaxine and Cytarabine
Number analyzed (Participants) | 36
Months | 3.1 [0.2 to 66.9]

4. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause
Time Frame: as for outcome 2
Measure: Median (Full Range); unit: Months
Arm/Group | Omacetaxine and Cytarabine
Number analyzed (Participants) | 36
Months | 8.1 [0.2 to 66.9]

5. Secondary Outcome: Induction Mortality
Description: Death within 8 weeks from the start of treatment.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Omacetaxine and Cytarabine
Number analyzed (Participants) | 36
Participants | 4

ADVERSE EVENTS:
Arm/Group | Omacetaxine and Cytarabine
All-Cause Mortality (participants affected / at risk) | 4/36
Serious Adverse Events (participants affected / at risk) | 20/36
Other Adverse Events (participants affected / at risk) | 15/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omacetaxine and Cytarabine (N=36)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Heart Failure (Cardiac disorders) | 1 (1)
Scleral Disorder (Eye disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Rectal Bleeding (Gastrointestinal disorders) | 1 (1)
Back Pain (General disorders) | 1 (1)
Death (General disorders) | 3 (3)
Fall (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Cholecystitis (Infections and infestations) | 1 (1)
Fever/Infection and Infestation (Infections and infestations) | 1 (1)
Joint Infection (Infections and infestations) | 1 (1)
Lung Infection (Infections and infestations) | 2 (2)
Neutropenic Fever (Infections and infestations) | 9 (12)
Sepsis (Infections and infestations) | 3 (3)
Sinusitis (Infections and infestations) | 1 (1)
Alanine Aminotransferase increased (Metabolism and nutrition disorders) | 1 (1)
Aspartate Aminotransferase increase (Metabolism and nutrition disorders) | 1 (1)
Creatinine increase (Metabolism and nutrition disorders) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleuritic pain (General disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omacetaxine and Cytarabine (N=36)
Alanine Aminotransferase increased (Metabolism and nutrition disorders) | 2 (2)
Asparatate Aminotransferase increase (Metabolism and nutrition disorders) | 2 (2)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 2 (2)
Neutropenic Fever (Infections and infestations) | 7 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (5)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes